CLINICAL TRIAL: NCT04947527
Title: Phase 2 Efficacy & Safety Evaluation of Advantage Anti-Caries Varnish for Primary Prevention
Brief Title: Efficacy and Safety Evaluation of Anti-Caries Varnish
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advantage Silver Dental Arrest, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019-10-19
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2024-08

CONDITIONS: Dental Caries in Children
Keywords: sodium fluoride; povidone iodine; dental varnish; primary dentition

STUDY DESIGN:
Intervention Model Description: This is a single center randomized, double-blind, placebo-controlled, parallel-group trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study personnel except for designated personnel in the data center will be blinded to the participant treatment assignment. In order to maintain blinding and eliminate examiner bias, the staff member applying these varnishes will not perform the caries scoring exams.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test Varnish (Experimental): Anti-Caries Varnish. The active ingredients are 10% (w/v) Povidone-Iodine and 5% (w/v) Sodium Fluoride CAS.
  Interventions: Drug: Test varnish
- Control Varnish (Active Comparator): Control Varnish. 5% (w/v) Sodium Fluoride .
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Test varnish — A maximum of 0.2 mL will be applied to the teeth with a dental brush. Test or control varnish will be applied topically 4 times per year following enrollment and at each 3 to 4-month intervals.
  Other Names: Advantage Anti-Caries Varnish
  Arms: Test Varnish
Drug: Placebo — A maximum of 0.2 mL will be applied to the teeth with a dental brush. Test or control varnish will be applied topically 4 times per year following enrollment and at each 3 to 4-month intervals.
  Other Names: Placebo Varnish; Fluoride Varnish
  Arms: Control Varnish

SUMMARY:
The purpose of the study is to determine the efficacy & safety of Advantage Anti-Caries Varnish for primary prevention. The objectives are:

1) To determine if Advantage Anti-Caries Varnish (test varnish) is superior to an active control varnish (5% Sodium Fluoride, no Povidone-Iodine) in the prevention of caries lesions in the primary dentition. Specifically, prevention of caries lesions in primary teeth that either are sound, have only d1 (white spots) lesions or unerupted at baseline; and 2) To document the safety of the test varnish.

DETAILED DESCRIPTION:
This is a single center randomized, double-blind, placebo-controlled, parallel-group trial. The treatment group will be exposed at baseline and once every three to four months after baseline for a maximum period of 24 months. The control group will be exposed to the control varnish in the same manner. 254 subjects will be enrolled. Half will be randomized to each arm. Subjects will be 6-24 mo of age and in good health. Children attending Maternal and Child Health (MCH) Immunization and Well Child programs in Pohnpei State will be enrolled. Primary Outcome Variables: 1) Surface-level dental caries lesions (d2-4mfs) at 24 months post baseline; 2) Presence/Absence of dental caries lesions (d2-4mfs >0) at 12 months post baseline. Secondary Outcome Variable: Adverse Events

ELIGIBILITY:
Inclusion Criteria:

1. The subject's parent or legal guardian must provide signed and dated informed consent (parent permission form).
2. The subject's parent or legal guardian of the subject must be willing and able to comply with study requirements.
3. The subject is a 6-24 months at the time of enrollment.
4. The subject must be in good general health as evidenced by parent report.
5. The subject will have at least 1 erupted tooth that is either sound or has only a d1 (white spots) lesion.

Exclusion Criteria:

1. Previous treatment with fluoride varnish
2. Known allergy to iodine
3. Diagnosis of thyroid disease
4. Chronic, prophylactic use of antibiotics
5. Treatment with another investigational drug or intervention within 30 days preceding the Baseline Visit.
6. Visible cavities (d2-4)
7. Presence of intraoral pathology that would make assessment of post treatment soft tissue ulcerations or inflammation impossible (child could be enrolled if problem is treated and lesions cleared)
8. Parent anticipates the child will move from Pohnpei during the next 2 years.

Ages: 10 Months to 20 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 274 (Actual)
Dates: Start 2022-06-04 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ohnmar K Tut, BDS Phil, Principal Investigator — University of Washington
Locations (1):
- Pohnpei State Hospital, Pohnpei, FSM, United States Minor Outlying Islands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Varnish | Control Varnish
Started | 132 | 142
Completed | 121 | 123
Not Completed | 11 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Varnish | Control Varnish | Total
Number analyzed (Participants) | 132 | 142 | 274
Age, Continuous [Mean (Standard Deviation); unit: Months] | 13.9 (4.4) | 14.3 (4.5) | 14.1 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 83 | 149
  Male | 66 | 59 | 125
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 132 | 142 | 274
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Caries Increment
Description: Surface-level dental caries lesions (d2-4mfs) at 24 months post baseline, which is the number of surfaces at 24 months post baseline with cavitation into the enamel (d2), dentin (d3) or pulp (d4), missing due to caries (m) or filled (f).
Time Frame: 24 months post baseline
Population: All children with follow-up at 24 months post-baseline.
Measure: Mean (Standard Deviation); unit: Number of tooth surfaces
Arm/Group | Test Varnish | Control Varnish
Number analyzed (Participants) | 121 | 123
Number of tooth surfaces | 9.8 (10.6) | 11.3 (10.8)
Statistical Analysis 1: Comparison: Test Varnish vs Control Varnish; Test type: Superiority; p = 0.279, t-test, 2 sided; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-4.2 to 1.2]

2. Primary Outcome: Number of Participants With Caries, Surfaces Missing Due to Caries or Filled Surfaces
Description: Presence/Absence of dental caries lesions (d2-4mfs >0), which is defined by the presence at 12 months post baseline of 1 or more tooth surfaces with cavitation into the enamel (d2), into the dentin (d3), or into the pulp (d4), missing due to caries (m) or filled (f).
Time Frame: 12 months post baseline
Population: All children with follow-up 12 months post-baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Test Varnish | Control Varnish
Number analyzed (Participants) | 124 | 126
Participants | 53 | 72
Statistical Analysis 1: Comparison: Test Varnish vs Control Varnish; Test type: Superiority; p = 0.023, Chi-squared; Difference in percentages/proportions = -14.4, 95% CI 2-sided [-26.7 to -2.1]

3. Secondary Outcome: Adverse Events
Description: Cumulative Adverse and Serious Adverse Events
Time Frame: 24 months post baseline
Measure: Count of Participants; unit: Participants
Groups:
- Test Varnish: Anti-Caries Varnish: The active ingredients are 10% (w/v) Povidone-Iodine and 5% (w/v) Sodium Fluoride CAS.
- Control Varnish: Control Varnish: 5% (w/v) Sodium Fluoride.
Arm/Group | Test Varnish | Control Varnish
Number analyzed (Participants) | 132 | 142
Participants | 42 | 58
Statistical Analysis 1: Comparison: Test Varnish vs Control Varnish; Test type: Superiority; p = 0.133, Fisher Exact; Risk Difference (RD) = -0.09

ADVERSE EVENTS:
Time Frame: Two years from baseline through 24-month follow-up.
Description: Primary collection approach was non-systematic by parent self-report, and secondary collection approach was systematic by dental exam at 12-month and 24-month follow-ups.
Arm/Group | Test Varnish | Control Varnish
All-Cause Mortality (participants affected / at risk) | 0/132 | 0/142
Serious Adverse Events (participants affected / at risk) | 0/132 | 0/142
Other Adverse Events (participants affected / at risk) | 42/132 | 58/142
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Varnish (N=132) | Control Varnish (N=142)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Blood deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Candidiasis (General disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 7 (7) | 11 (11)
Flu (Infections and infestations) | 31 (36) | 44 (47)
Pink eye (Infections and infestations) | 0 (0) | 1 (1)
Runny nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin rash (Immune system disorders) | 0 (0) | 1 (1)
Small vesicles (Immune system disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT04947527/Prot_SAP_000.pdf